CLINICAL TRIAL: NCT02955849
Title: The China Laser and Surgery Study : A Mixed Methods Study With an Random Control Trial Comparing Outcomes From Selective Laser Trabeculoplasty Versus Surgical Treatment (Trabeculectomy) for Glaucoma in Rural China .
Brief Title: A Trial of China Laser and Surgery Study Glaucoma in Rural China
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, vice directior, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLT in rural China
Record Dates: First submitted 2016-04-11; First posted 2016-11-04 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: glaucoma; rural; China; SLT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SLT laser group (Experimental): 1. selective laser trabeculoplasty for 360 degrees the study eye.
  2. Patients having 1 or 2 quadrants of angle with trabecular meshwork not visible will undergo Laser peripheral iridotomy prior to selective laser trabeculoplasty to maximize the amount of angle visible;
  3. Cataract surgery will be offered if indicated and completed within 3 months of selective laser trabeculoplasty , if accepted by the patient.
  4. Patients will be re-examined every 4 months and selective laser trabeculoplasty performed again according to the above protocol if intraocular pressure exceeds the target (25% reduction from the original intraocular pressure or < 21 mmHg, whichever is lower).
  Interventions: Device: SLT laser
- Standard care group (No Intervention): * Trabeculectomy as usually performed by the operative surgeon in one eye (study eye).
  * Both Mitomycin and releasable sutures are permitted if indicated in the opinion of the surgeon and s/he can perform and/or has access.
  * Simultaneous cataract surgery is permitted if indicated in the opinion of the operating surgeon.
  * Patients will be re-examined every 4 months， and Timolol 0.5% added bid if intraocular pressure exceeds the target (25% reduction from the original intraocular pressure or < 21 mmHg, whichever is lower)
- Drug treatment group (No Intervention): Patients not accepting the offered treatment for the study eye within 3 months will receive topical Timolol 0.5% bid at the usual price, with the prescription to be refilled per usual practice at the hospital (usually monthly).

INTERVENTIONS:
Device: SLT laser — Patients will be offered initial SLT laser by doctors
  Arms: SLT laser group

SUMMARY:
Aims and Objectives (Quantitative) Aim: To compare the effectiveness of selective laser trabeculoplasty with trabeculoplasty in lowering the intraocular pressure in patients with medically uncontrolled open angle glaucoma in rural China, taking into account the impact of patient acceptance of each type of treatment

Hypothesis: Mean intraocular pressure after treatment with selective laser trabeculoplasty will be lower than with surgery due to higher acceptance rates among patients randomized to receive this treatment and therefore treatment provided at an earlier stage of disease progression.

DETAILED DESCRIPTION:
Glaucoma is one of the three leading causes of blindness in China. Although this condition can be controlled with medication to lower intraocular pressure , such treatment must continue over a patient's lifetime. This is not practical in resource-poor settings due to cost and inconvenience for patients. Trabeculectomy is the standard treatment offered in rural China but is rarely used because of the following issues:

1. need for hospitalization, which increases patient expense and inconvenience
2. high refusal rates by patients for all ocular surgery
3. high rates of infection due to poor quality instruments and material
4. need for multiple follow-up visits post-surgery (our earlier work shows a return rate of only 30% 1 month post-surgery among rural patients in China).

A viable alternative for patients in rural China is selective laser trabeculoplasty , based on the following advantages:

1. simplicity (done as a 5-minute out-patient procedure requiring only topical anaesthesia)
2. effectiveness (18-32% reduction in intraocular pressure, which is comparable to medication)
3. safety (complications are rare and do not include serious infectious as with trabeculotemy)
4. convenience (minimal follow-up, with one visit within 6 weeks post-surgery)
5. cost-effectiveness (compared to other glaucoma therapies in many settings)
6. acceptability to patients (due to low-cost out-patient care with easy follow-up).

Study Design (Quantitative) This phase of the proposed China Laser and Surgery Study research project is a multi-centre open-label pragmatic randomised controlled trial.

Expected timeline:

* Enrolment: 12 months
* Follow-up: 12 months
* Data analysis: 4 months

Patient Population and Setting: Patients presenting with glaucoma at rural hospitals (n=4) in Guangdong province, China, all of whom are currently capable of performing trabeculectomy surgery, and have been provided an selective laser trabeculoplasty machine and training in its use.

Sample Size: One hundred ninety patients (95 in each group) will be needed to obtain a power of 0.90, with a two-sided alpha of 0.05. Patients are the unit of randomization. Expected IOP difference between groups of 3.0 mm Hg + 4.0 mmg HG, and a correlation of 0.30 between baseline and final intraocular pressure, allowing for loss to follow up of 30%.

Baseline Data:

aseline data (to be collected prior to determination of eligibility and randomization but after obtaining informed consent) include the following:

* Presence or absence of relevant pre-existing health conditions (i.e., hypertension, diabetes, cardiovascular disease)
* Ophthamologic test results

  * Best corrected visual acuity and presenting visual acuity in both eyes
  * Intraocular pressure in both eyes
  * Cup to disk ratio in both eyes
  * presence or absence of visually significant cataract in both eyes; if cataract present in study eye, whether cataract surgery has already been performed
  * degrees of visible Trabecular Meshwork in the study eye on gonioscopy without "dynamic gonioscopy"
* score on glaucoma knowledge test using a simple, previously validated questionnaire
* Demographic data

  * date of birth or self-reported age in years
  * sex
* Contact information

  * Address
  * mobile phone number where can be reached (own or neighbours, etc.)
* Socioeconomic status

  * completed education in years
  * wealth, as measured by ownership of items on a pre-determined list of 13 common household devices in China
  * job title/description
* Level of difficulty traveling to hospital with eye clinic

  * distance traveled
  * time spent traveling
  * direct or out-of-pocket costs for travel, meals, etc.

Main analyses:

* Following requirements for intention-to-treat analyses, we will measure mean intraocular pressure at 12 months comparing the two groups and adjusting for baseline intraocular pressure, including all subjects who accepted and refused treatment (primary analysis, unadjusted). We will also measure intraocular pressure as above, adjusting for cataract surgery, age, gender, prior use of medication, degrees of open angle in study eye at baseline, and severity of glaucoma (Cup to disk ratio) in study eye at baseline (primary analysis, adjusted). Both of the above analyses will be repeated using a per protocol approach (including only patients who accepted their assigned therapy, or secondary analysis).
* We will test for differences in baseline characteristics by study group with t-tests (for continuous variables) and Chi-square tests (for categorical variables). We will use generalized linear models with Poisson regression (for variables with binary outcomes) and linear regression (for variables with continuous outcomes) to estimate the relative risk for the intervention arm. Multiple imputation in Stata 13.1 (StataCorp, College Station, TX, USA) will be used to address missing data. All statistical analysis will be performed using Stata 13.1. A two-tailed P-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of glaucoma (Cup to disk ratio, or CDR > 0.6 with optic nerve appearance and/or visual field findings consistent with glaucoma in the study eye)
* angle configuration > 180° of trabecular meshwork visible in the study eye
* no previous ocular incisional surgery or ocular laser treatment except refractive or cataract surgery in the study eye
* Best corrected visual acuity > 6/60 metres in both eyes

Exclusion Criteria:

* Intraocular pressure > 35 in the study eye
* Cup to disk ratio > 0.9 in the study eye
* Inability to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 12 months
  * intraocular pressure in study eye 12 months after receiving treatment (laser or surgery)
  * the intraocular pressure of patients refusing their allocated intervention will still be recorded at 12 months post-refusal and will be considered in the analysis
  * patients accepting the allocated treatment > 3 months after initial offer of treatment will be considered as having refused and their outcome intraocular pressure will be the last reading prior to treatment

SECONDARY OUTCOMES:
Visual quality of life | 12 months
  use the scale "NEI-VQ 25" to assess the patient's visual quality of life
Satisfaction score | 12 months
  Using a Surgical Satisfaction Questionnaire previously validated in rural China
Cataract surgery | 12 months
  Cataract surgery performed in conjunction with allocated treatment (Yes/No)
Allocated treatment | 12 months
  use acceptance questionnaire form to calculate surgical receiving rate

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD,MPH, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Blindness Preventment and Treatment Department, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Liang YB, Friedman DS, Wong TY, Zhan SY, Sun LP, Wang JJ, Duan XR, Yang XH, Wang FH, Zhou Q, Wang NL; Handan Eye Study Group. Prevalence and causes of low vision and blindness in a rural chinese adult population: the Handan Eye Study. Ophthalmology. 2008 Nov;115(11):1965-72. doi: 10.1016/j.ophtha.2008.05.030. Epub 2008 Aug 5. PMID 18684506
- [Background] Zhang XJ, Liang YB, Liu YP, Jhanji V, Musch DC, Peng Y, Zheng CR, Zhang HX, Chen P, Tang X, Lam DS. Implementation of a free cataract surgery program in rural China: a community-based randomized interventional study. Ophthalmology. 2013 Feb;120(2):260-5. doi: 10.1016/j.ophtha.2012.07.087. Epub 2012 Oct 27. PMID 23107580
- [Background] Ang GS, Varga Z, Shaarawy T. Postoperative infection in penetrating versus non-penetrating glaucoma surgery. Br J Ophthalmol. 2010 Dec;94(12):1571-6. doi: 10.1136/bjo.2009.163923. Epub 2009 Nov 5. PMID 19897472
- [Background] Liu T, Congdon N, Yan X, Jin L, Wu Y, Friedman D, He M. A randomized, controlled trial of an intervention promoting cataract surgery acceptance in rural China: the Guangzhou Uptake of Surgery Trial (GUSTO). Invest Ophthalmol Vis Sci. 2012 Aug 13;53(9):5271-8. doi: 10.1167/iovs.12-9798. PMID 22789919
- [Background] Wittenborn JS, Rein DB. Cost-effectiveness of glaucoma interventions in Barbados and Ghana. Optom Vis Sci. 2011 Jan;88(1):155-63. doi: 10.1097/OPX.0b013e3181fc30f3. PMID 21076360
- [Background] Narayanaswamy A, Leung CK, Istiantoro DV, Perera SA, Ho CL, Nongpiur ME, Baskaran M, Htoon HM, Wong TT, Goh D, Su DH, Belkin M, Aung T. Efficacy of selective laser trabeculoplasty in primary angle-closure glaucoma: a randomized clinical trial. JAMA Ophthalmol. 2015 Feb;133(2):206-12. doi: 10.1001/jamaophthalmol.2014.4893. PMID 25429421
- [Background] Realini T. Selective laser trabeculoplasty for the management of open-angle glaucoma in St. Lucia. JAMA Ophthalmol. 2013 Mar;131(3):321-7. doi: 10.1001/jamaophthalmol.2013.1706. PMID 23348420
- [Background] Adekoya BJ, Akinsola FB, Balogun BG, Balogun MM, Ibidapo OO. Patient refusal of glaucoma surgery and associated factors in Lagos, Nigeria. Middle East Afr J Ophthalmol. 2013 Apr-Jun;20(2):168-73. doi: 10.4103/0974-9233.110612. PMID 23741137